CLINICAL TRIAL: NCT01007565
Title: Postoperative Pain After Volar Plating for Distal Radius Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-0801/053-013
Record Dates: First submitted 2009-11-01; First posted 2009-11-04 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Distal Radius Fractures
Keywords: periarticular injection
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- periarticular injection, pain level (Experimental)
  Interventions: Procedure: periarticular anesthetics injection

INTERVENTIONS:
Procedure: periarticular anesthetics injection — Members in the PI group received intra-operative periarticular injections and additional sensory nerve blocks just before skin closure . For the periarticular injections and additional sensory block, local analgesic solution was injected into the wrist joint, joint capsule, periosteum, subcutaneous tissue, skin, and around the anterior and posterior interosseous nerves and the superficial radial nerve. A volume of 2ml was injected into the joint capsule and periosteum, and of 3ml into the wrist joint, subcutaneous tissue, skin and into each nerve.

SUMMARY:
The investigators undertook to evaluate early postoperative pain levels after the volar plating of distal radius fractures performed under regional anesthesia, and to determine whether periarticular multimodal drug injections into the joint, ligament, periosteum, subcutaneous tissue, and skin, and into interosseous and superficial radial nerves (as an additional sensory nerve block) provide additional pain management benefits.

DETAILED DESCRIPTION:
To evaluate whether periarticular injections (PI) had additional pain management benefits, patients were randomly allocated to two groups, that is, the PI and No-PI groups, using a randomization table. Members in the PI group received intra-operative periarticular injections and additional sensory nerve blocks just before skin closure. For the periarticular injections and additional sensory block, local analgesic solution was injected into the wrist joint, joint capsule, periosteum, subcutaneous tissue, skin, and around the anterior and posterior interosseous nerves and the superficial radial nerve.

A volume of 2ml was injected into the joint capsule and periosteum, and of 3ml into the wrist joint, subcutaneous tissue, skin and into each nerve. The anterior interosseous nerve was blocked in the course of the pronator quadratus and posterior interosseous nerve in the 4th dorsal extensor compartment.

The mixture of anesthetics consisted of 2 ampules of ropivacaine HCl (Naropin®, 0.75%, 7.5mg/ml, 20ml/ⓐ), 1 ampule of morphine sulfate (5mg/ⓐ), 1 ampule of epinephrine HCL (1mg/ml, 1ml/ⓐ) and normal saline 20cc.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture with or without a styloid fracture not requiring surgery

Exclusion Criteria:

* multiple trauma
* a combined distal radio-ulnar joint instability or a large ulnar styloid fragment requiring fixation
* regularly narcotics user
* those with a psychiatric illness, a major systemic illness or a known allergy or contraindication to opiates or local anesthetics.

Ages: 16 Years to 89 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
postoperative pain level | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Sik Gong, Professor, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of orthopedic surgery, Seoul national university bundang hospital, Seongnam-si, Gyeonggi-do, South Korea